CLINICAL TRIAL: NCT04395534
Title: Non-microradical Resection Margin as a Predictor for Recurrence After Complete Mesocolic Excision: a Prospective Cohort Study
Brief Title: Non-microradical Resection Margin as a Predictor for Recurrence After Complete Mesocolic Excision
Status: Completed | Type: Observational
Sponsor: Claus Anders Bertelsen, PhD, MD (Other)
Responsible Party: Sponsor-Investigator, Claus Anders Bertelsen, PhD, MD, Consultant Colorectal Surgeon, Associate Professor, Head of Research Department of Surgery, Nordsjaellands Hospital
Organization: Nordsjaellands Hospital (Other)
Other Study IDs: R1 - CME
Record Dates: First submitted 2020-05-15; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Complete mesocolic excision

SUMMARY:
The study aim to investigate the value of the current definition of microradical resection margin in colon cancer. Is the distance from tumor tissue to resection margin and the site of any clinically prognostic importance if complete mesocolic excision has been performed.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective curative intended complete mesocolic excision for primary colon adenocarcinoma at Nordsjællands Hospital in Hillerød, Denmark
* International Union Against Cancer (Union Internationale Contre le Cancer - UICC) stage III - pT1-4, pN1-2 cM0 (gastroepiploic and infrapyloric lymph node metastases are not considered as distant metastases)
* Resident in Denmark at the time of surgery.

Exclusion Criteria:

* Patients who did not undergo macroradical resections
* Synchronous colorectal cancer
* Venous invasion at central venous ligation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective curative intended complete mesocolic excision for primary colon adenocarcinoma at Nordsjællands Hospital in Hillerød, Denmark
Sampling Method: Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2008-06-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Recurrence | 3 years
  Any type of recurrence

REFERENCES:
- [Derived] Gundestrup AK, Olsen ASF, Ingeholm P, Bols B, Kleif J, Bertelsen CA. Nonmicroradical Resection Margin as a Predictor of Recurrence in Patients With Stage III Colon Cancer Undergoing Complete Mesocolic Excision: A Prospective Cohort Study. Dis Colon Rectum. 2022 May 1;65(5):683-691. doi: 10.1097/DCR.0000000000001996. PMID 34933419